CLINICAL TRIAL: NCT05448547
Title: A Randomized, Open-label, Multicenter, Parallel Group Treatment, Phase 3, Two-arm Study to Measure the Effect on Overall Survival and Quality of Life of Immediate Curative Therapy Compared With Standard Conservative Treatment in Older Male Participants Aged ≥ 75 Years With Non-metastatic, High-risk Prostate Cancer
Brief Title: Immediate Curative vs Conservative Treatment in Older Men With M0, High-risk Prostate Cancer
Acronym: GrandP/SPCG19
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sven Löffeler (Other)
Collaborators: Oslo University Hospital (Other); Klinbeforsk (Other)
Responsible Party: Sponsor-Investigator, Sven Löffeler, Principal investigator, The Hospital of Vestfold
Organization: The Hospital of Vestfold (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GrandP
Record Dates: First submitted 2022-06-22; First posted 2022-07-07 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; older patients; immediate curative treatment; conservative treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: randomized, parallel, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate curative therapy (Experimental): Patients randomized to the intervention arm will receive immediate curative therapy in the form of either radiotherapy to the prostate in combination with hormone therapy (ADT or monotherapy) or surgery (radical prostatectomy). Standard treatment in this arm is radiotherapy + hormone therapy. Surgery is reserved for patients with strong preferences against radiotherapy.
  Interventions: Radiation: Radiotherapy or surgery
- initial observation/ hormone therapy (Active Comparator): Patients in this arm will either be observed (with localized high-risk prostate cancer) or receive hormone therapy (locally advanced prostate cancer; ADT or monotherapy). Further local or systemic therapy is given at doctor's discretion triggered by local or/ and systemic progression.
  Interventions: Other: initial observation; Drug: Hormone therapy

INTERVENTIONS:
Radiation: Radiotherapy or surgery — see arm/ group description
  Arms: immediate curative therapy
Other: initial observation — see arm/ group description
  Arms: initial observation/ hormone therapy
Drug: Hormone therapy — androgen depression therapy (ADT) by either LHRH agonist or antagonist or androgen monotherapy
  Arms: initial observation/ hormone therapy

SUMMARY:
It is currently unclear if immediate curative treatment (radiotherapy or surgery) of high-risk prostate cancer without metastasis in older men (>=75 years) generates the same survival benefits as in younger patients or if the harms/ side-effects of immediate curative treatment outweigh the benefits. In this study the investigators randomize older patients with high-risk, non-metastatic high-risk prostate cancer to either immediate curative therapy or to conservative, more problem-oriented therapy to investigate if immediate curative treatment prolongs life, improves quality of life and is cost-effective.

DETAILED DESCRIPTION:
There is a lack of both level 1 evidence and consensus regarding the optimal treatment strategy for older men (>=75 years) with non-metastatic, high-risk prostate cancer. Currently, in Scandinavia, the majority of older patients are treated conservatively, i.e. with hormone therapy or watchful waiting while some centers recommend immediate curative therapy regardless of patient age. Older patients thus risk both undertreatment and overtreatment of their cancer. This randomized clinical trial investigates if immediate curative therapy of high-risk, non-metastatic prostate cancer prolongs life (as it does in younger patients) and improves health-related quality of life. Furthermore, this trial investigates if the early side effects of immediate curative therapy are compensated by better long-term tumor control, better quality of life, functional status and improved survival.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 75 years of age or older, at the time of signing the informed consent.
2. Participants who are healthy as determined by medical evaluation and geriatric G8/ miniCOGTM evaluation (G8: Fit, score >14, or reversibly frail; miniCOGTM: score >2)

   And who have PCa (diagnosed ≤6 months) with one or both of the following features:
   * Gleason grade 8-10 (ISUP group 4 and 5) other than microscopic, low-volume disease (tumor must be either palpable or visible on MRI, i.e., PIRADS 4 or 5)
   * Locally advanced PCa (T3 or T4) (unequivocal findings of clinical/ radiological T3 or clinical/ radiological T4 on DRE or MRI; broad capsular contact of tumor on MRI is treated as localized disease, T2, in the context of this study)
   * Able to read, understand and fill in HRQoL questionnaires (PROMS)
3. Male
4. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Medical Conditions

1. Dementia (unable to consent) Prior/Concomitant Therapy
2. Prior radiation to the pelvis
3. Hormone therapy >3 months prior to randomization Diagnostic assessments
4. Lymph node metastasis (N0) on MRI, CT or PSMA-PET CT (equivocal N-findings =N0; borderline cases will be discussed and called by a study tumor board).
5. Distant metastasis (M0) on MRI, CT, bone scan or PSMA-PET CT (equivocal bone scan findings need to be confirmed with MRI or CT; borderline cases will be discussed by a study tumor board).

   Other Exclusions
6. Disabled or severe comorbidity (identified by G8 screening)
7. Unable to read, understand or fill out HRQoL questionnaires (PROMS)

Min Age: 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Only males have prostate cancer
Enrollment: 980 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years following end of recruitment
  overall survival
Burden of disease | 0-10 years
  European Organisation for Research and Treatment of Cancer questionnaire for assessment of health-related quality of life elderly patients with cancer (EORTC ELD 14), burden of disease scale (2 questions, score 0-100, high scores indicate high burden of disease)

SECONDARY OUTCOMES:
Role functioning | 0-10 years
  European Organisation for Research and Treatment of Cancer questionnaire for quality of life of cancer patients (EORTC-QLQ-C30), RF2 scale (2 questions, score 0-100, high scores indicate a high / healthy level of functioning)
Urinary irritative/ obstructive symptoms | 0-10 years
  Expanded Prostate Cancer Index Composite Short Form questionnaire (EPIC-26),urinary scales (score 0-100, higher scores indicating better outcomes)
bowel symptoms | 0-10 years
  Expanded Prostate Cancer Index Composite Short Form questionnaire (EPIC-26), bowel scales (score 0-100, higher scores indicating better outcomes)
Prostate cancer morbidity | 0-10 years
  hospitalizations, interventions, complications due to local progression/ systemic progression)
Prostate-cancer-specific survival | 0-10 years
  Prostate cancer deaths in intervention and control group
Metastasis-free survival | 0-10 years
  time to metastasis detected radiographically due to symptoms or biochemical progression
Symptom-/ intervention-free survival | 0-10 years
  time to symptoms/ need for interventions due to prostate cancer progression
Quality of life-adjusted years | 0-10 years
  Euro QoL group questionaire (EQ-5D-5L) (1 =full health; 0= dead)
need for secondary and tertiary therapy | 0-10 years
  use of second- and third-line therapies

OTHER OUTCOMES:
Institutionalized care | 0-10 years
  at each follow-up visit the living status of the patients will be assessed. If patients have become dependent on permanent nursing home/ assisted care this will be registered.
Health-related quality of life in cancer patients | 0-10 years
  European Organisation for Research and Treatment of Cancer questionnaire for quality of life of cancer patients (EORTC-QLQ-C30), scales not primary/ secondary outcome measures (All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems)
Health-related quality of life in older cancer patients | 0-10 years
  European Organisation for Research and Treatment of Cancer questionnaire for quality of life of cancer patients (EORTC-QLQ-C30), scales not primary outcome (All of the scales and single-item measures range in score from 0 to 100. High scores indicate poor mobility, good family support, much worry about the future, good maintenance of autonomy and purpose)
Quality of Life issues in patients with prostate cancer | 0-10 years
  Expanded Prostate Cancer Index Composite Short Form questionnaire (EPIC-26), scales not secondary outcomes (score 0-100, higher scores indicating better outcomes)
Instrumental activities of daily living (iADL) | 0-10 years
  Lawton and Brody questionnaire (8 questions, minimum score 0, maximum score 5, higher scores indicating need for assistance)
Personal activities of daily living (pADL) | 0-10 years
  Lawton and Brody questionnaire (6 questions, minimum score 0, maximum score 5, higher scores indicating need for assistance)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Loffeler, MD, PhD, Principal Investigator — The Hospital of Vestfold
Locations (18):
- Denmark (3):
  - Rigshospital, Copenhagen
  - Esbjerg and Grindsted Hospital, Esbjerg
  - Odense University Hospital, Odense
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Norway (11):
  - Sunmøre Hospital Trust, Ålesund, Møre og Romsdal
  - Oslo University Hospital, Oslo, Oslo County
  - Stavanger University Hospital, Stavanger, Rogaland
  - Sørlandet Hospital Trust, Kristiansand, Sørlandet
  - Telemark Hospital Trust, Skien, Telemark
  - St. Olavs Hospital, Trondheim, Trøndelag
  - Vestfold Hospital Trust (Hospital of Vestfold), Tønsberg, Vestfold
  - Vestre Viken Hospital Trust, Drammen
  - Innlandet Hospital Trust, Hamar
  - Akerhus University Hospital, Lørenskog
  - University Hospital of Northern Norway, Tromsø
- Capio Saint Göran's Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Only anonymized data will be shared

REFERENCES:
- [Derived] Loffeler S, Bertilsson H, Muller C, Aas K, Haugnes HS, Aksnessaether B, Pesonen M, Thon K, Tandstad T, Murtola T, Poulsen MH, Nordstrom T, Vigmostad MN, Ottosson F, Holmsten K, Christiansen O, Slaaen M, Haug ES, Storas AH, Asphaug L, Rannikko A, Brasso K; Scandinavian Prostate Cancer Group (SPCG) and the Norwegian Get-Randomized (GRand) Initiative. Protocol of a randomised, controlled trial comparing immediate curative therapy with conservative treatment in men aged >/=75 years with non-metastatic high-risk prostate cancer (SPCG 19/GRand-P). BJU Int. 2024 Jun;133(6):680-689. doi: 10.1111/bju.16314. Epub 2024 Mar 12. PMID 38469686